CLINICAL TRIAL: NCT05858944
Title: Home Blood Pressure Intervention in the Community Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Hypertension (Other)
Responsible Party: Principal Investigator, Yan Li, Professor, Doctor of Medicine, Doctor of Philosophy, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.1
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Home Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive Home BP Control (Experimental): Participants randomized into the intensive treatment arm will have a goal of home BP<125/75 mmHg.
  Interventions: Drug: Intensive Home BP control
- Standard Home BP Control (Active Comparator): Participants randomized into the standard treatment arm will have a goal of home BP within 125-134/75-84 mmHg.
  Interventions: Drug: Standard Home BP control

INTERVENTIONS:
Drug: Intensive Home BP control — If the target home BP level is not achieved during the follow-up periods, type and dosage of antihypertensive drugs will be adjusted according to current guidelines and physician's clinical experience.
  Other Names: Home BP<125/75 mmHg
  Arms: Intensive Home BP Control
Drug: Standard Home BP control — If the target home BP level is not achieved during the follow-up periods, type and dosage of antihypertensive drugs will be adjusted according to current guidelines and physician's clinical experience.
  Other Names: Home BP<135/85 mmHg
  Arms: Standard Home BP Control

SUMMARY:
The primary purpose of the study is to explore whether a lower home blood pressure target (125/75 v.s. 135/85 mmHg) would be beneficial to elderly treated hypertensive patients in terms of reduced incidence of cardiovascular events. The study also aims to promote the application of standardised and information-based home blood pressure monitoring in community hypertension management.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 years old
* Have been taking antihypertensive drugs for more than 2 weeks
* The average SBP and/or DBP of 7-day home blood pressure monitoring ≥135/85 mmHg
* Willing to participate, adhere to follow-up, and sign the written informed consent form

Exclusion Criteria:

* Arm circumference too large or too small (less than 18 cm or greater than 42 cm) to fit the cuff in case of inaccurate measurement
* Invalid home blood pressure monitoring. The valid home blood pressure monitoring requires consecutive measurements for at least 3 days, with not less than 1 measurement in the morning and evening, respectively.
* Office blood pressure indicates stage 3 clinic hypertension (≥180/110 mmHg) during the screening period
* Suspected or known secondary hypertension
* Orthostatic hypotension, defined as a decrease in systolic blood pressure greater than 20 mmHg or diastolic blood pressure greater than 10 mmHg within 3 minutes when position is changed from sitting to standing
* eGFR<30 ml/min/1.73m2 or end-stage renal disease
* Cardiovascular events occured within the past 3 months, such as myocardial infarction, stroke, acute heart failure, hospitalization for unstable angina, undergoing coronary artery revascularization or bypass grafting
* Abnormal liver function (ALT/AST/total bilirubin more than 2 times the upper limit of normal value)
* Severe somatic disease with a life expectancy of less than 3 years, or diagnosed with cancer within the past 2 years requiring treatment
* Doctors deem that the participation would do harm to the patients or the patients would have poor compliance.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of adverse cardiovascular events | 48 months
  Composite of major adverse cardiovascular events consisting of death from cardiovascular diseases, non-fatal stroke, myocardial infarction, coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]), hospitalization for heart failure or unstable agina.

SECONDARY OUTCOMES:
Components of the primary outcome | 48 months
  Occurrence of any components of the primary outcome (death from cardiovascular diseases, non-fatal stroke, myocardial infarction, coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]), hospitalization for heart failure or unstable agina).
Renal outcome | 48 months
  Including end stage renal disease (ESRD) and a decrease in the eGFR of 30% or more
Adverse or severe adverse events | 48 months
  Especially dizziness and falls caused by hypotension, and orthostatic hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Professor, Principal Investigator — Shanghai Institute of Hypertension; Jiguang Wang, Professor, Principal Investigator — Shanghai Institute of Hypertension
Locations (1):
- Community hospitals, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang DY, Zhang YQ, An DW, Cheng YB, Tang ST, Liu M, Li J, Staessen JA, Wang JG, Li Y; HomeBP Trial Investigators. A randomised trial comparing usual versus strict home blood pressure control in elderly patients with hypertension: protocol and initial progress. Blood Press. 2025 Dec;34(1):2472192. doi: 10.1080/08037051.2025.2472192. Epub 2025 Mar 2. PMID 39993302